CLINICAL TRIAL: NCT00030069
Title: Calcitriol and Dexamethasone for Myelodysplastic Syndromes
Brief Title: Calcitriol and Dexamethasone in Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Robert Redner, MD, Principal Investigator, University of Pittsburgh
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 01-020; FD-R-002025-01
Record Dates: First submitted 2002-01-30; First posted 2002-01-31 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: Hematopoiesis; Apoptosis; Cell Differentiation; Bone Marrow Cells
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Calcitriol; Dexamethasone

INTERVENTIONS:
Drug: Calcitriol
Drug: Dexamethasone

SUMMARY:
This is a study to determine the response rate in patients with myelodysplastic syndromes treated with calcitriol and dexamethasone.

DETAILED DESCRIPTION:
Current therapeutic options for myelodysplastic syndromes (MDS) are limited and, aside from bone marrow transplantation, none have proven superior to supportive measures alone. Preclinical investigations have indicated the potential therapeutic role for vitamin D in the treatment of MDS. However, because of the dose-limiting toxicity of hypercalcemia, past clinical trials with vitamin D have been forced to utilize low doses, with promising but inconsistent results.

This study utilizes a dosing schema of dexamethasone (Dex) and calcitriol (the active form of vitamin D) that augments the therapeutic index of calcitriol, and allows for safe administration of 5-10 times higher dose of calcitriol than previously has been used in clinical trials for MDS. Patients will receive dexamethasone 4 times per week and calcitriol 3 times per week. This schedule will continue weekly until patients are off study. The dose of calcitriol will be increased until the maximum tolerated dose (MTD) is determined. History and physical examination, blood monitoring, urinary ultrasounds, and bone marrow aspirations and biopsies will be used to assess disease response.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed refractory anemia (RA), RA with excess blasts (RAEB), RAEB in transformation (RAEB-IT), or ringed sideroblasts (RARS)
* Evidence of cytopenia affecting at least 1 hematological cell lineage
* Adequate liver and renal function
* ECOG 0-2
* Expected survival of at least 12 weeks

Exclusion criteria:

* Symptomatic coronary artery disease
* Uncontrolled diabetes mellitus
* Uncontrolled and symptomatic glaucoma
* History of dangerous reactions to steroid therapy
* Chemotherapy or any hematopoietic growth factor therapy within the past 8 weeks
* History of nephrolithiasis
* Children
* Chronic myelomonocytic leukemia (CMML)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2001-09; Primary Completion 2007-09 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States